CLINICAL TRIAL: NCT00794950
Title: A Phase II Study of Intravesical Bacillus Calmette-Guerin Followed by Sunitinib for the Treatment of High Risk Non-muscle Invasive Lower Urinary Tract Urothelial Carcinoma
Brief Title: Bacillus Calmette-Guerin Followed by Sunitinib for the Treatment of High Risk Non-muscle Invasive Lower Urinary Tract Urothelial Carcinoma
Acronym: Sutent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alon Weizer, Associate Professor Urology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sutent V5 / November 9, 2009
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Urinary Tract Urothelial Carcinoma
Keywords: Bladder Cancer; High Risk Non-muscle Invasive Lower Urinary Tract Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sunitinib treatment (Experimental): Intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients are treated with a 6-week induction course of intravesical bacillus Calmette-Guerin (BCG) followed by a 2 week rest period and 4 week course of oral Sunitinib.
  Patients will receive intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma. Two weeks after completion of BCG, patients will receive Sunitinib (50 mg daily) continuously for 28 days followed by a two week rest period. Patients will be reassessed with transurethral resection and urine cytology. Those with residual/recurrent disease will receive a second course identical to the initial protocol. Those with a complete response following initial or second treatment will be placed on maintenance BCG (3 week course every 6 months for 2 years). Those failing (progression, intolerance) initial/secondary treatments will be offered alternative therapy.
  Other Names: Sutent

SUMMARY:
A majority of patients with bladder cancer have disease confined to the inner lining of the bladder. Patients with high risk features (high grade tumors, tumors invading into a deeper superficial layer) are routinely treated with Bacillus Calmette Guerin (BCG) instilled in their bladder after the tumor has been removed. While up to 55% of patients respond to BCG, failure to respond may suggest a more aggressive tumor that requires more definitive therapy with complete bladder removal. BCG is believed to work by stimulating the body's own immune system to attack tumor cells. It may also work by blocking the machinery that tumors use to grow blood vessels which fuel tumor growth. A newer oral drug, sunitinib has shown to help patients with metastatic bladder cancer by blocking new blood vessel growth (VEGF inhibition). The investigators are studying the use of BCG followed by sunitinib in patients with high risk non-muscle invasive bladder cancer to evaluate the complete response (no visible evidence of tumor in the bladder) at 3 months and 6 months. The investigators will also evaluate whether there is recurrent tumor at three years.

DETAILED DESCRIPTION:
Despite a complete response of 45-55% in patients with non-muscle invasive urothelial carcinoma involving the lower urinary tract at 3 months, many patients suffer from multiple recurrences and progression in up to 1/3 of patients. While radical cystectomy is an effective local therapy for patients with high risk non-invasive disease, roughly 15% of patients will still develop progression. More importantly, the morbidity of radical cystectomy as described above represents a barrier to treatment in some individuals. Thus, there is a real need to identify newer therapies that reduce morbidity and improve outcomes in patients with non-invasive urothelial cancer. While multiple drug regimens have been the standard for many forms of cancer including invasive bladder cancer, few reports exist on multidrug regimens for non-invasive bladder cancer.

The fundamentally agreed upon mechanism of action of BCG intravesical therapy for superficial bladder cancer is the generation of a non-specific immune response with the expression of cytokines by inflammatory cells resulting in tumor death. Cytokines produced by BCG therapy such as IFNα may block vascular endothelial growth factor (VEGF) which is expressed in superficial and invasive bladder cancer and may provide a mechanism for disease progression.

Sunitinib is an oral tyrosine kinase inhibitor that blocks VEGF. Recent reports demonstrate clinical response in patients with metastatic bladder cancer treated with sunitinib after recurrence following standard chemotherapeutic regimens. The addition of sunitinib following BCG in order to consolidate VEGF inhibition may result in superior 3 month complete response rates. We know that patients who have a complete response to BCG at 3 months have improved disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed urothelial carcinoma confined to the urinary bladder and/or prostatic urethra by bladder biopsy within 6 weeks of study enrollment.
* Patients are eligible if the biopsy was done within 3 months of enrollment and a cystoscopy demonstrates no gross disease within 6 weeks of enrollment.
* Tumor histology with >50% transitional cell carcinoma histology
* Tumor stage less than or equal to T1 confirmed by pathology report
* Patients with a T1 tumor will require a restaging TURBT confirming no higher stage tumor prior to study enrollment
* High grade tumor as defined by the WHO/ISUP 1998 classification system. (Presence of carcinoma in situ constitutes a high grade tumor)
* No BCG within 12 months of enrollment
* Patients are allowed to have received a single dose of intravesical chemotherapy (excluding BCG) in the operating room following transurethral resection documenting non-muscle invasive urothelial carcinoma of the lower urinary tract.
* Patients are allowed to have received a previous 6 week cycle of any standard intravesical chemotherapy if > 3 months prior to enrollment.
* Age >18 years.
* ECOG performance status 0 or 1
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count > 1,500/mcL
  * platelets > 100,000/mcL
  * total bilirubin less than or equal to 1.5 upper limit of normal
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper
  * limit of normal
  * Serum creatinine < 2.0 mg/dl
  * MUGA scan within institutional normal limits
* Timing guideline for pre-study labs and measurements:
* All pre-study labs required for determination of eligibility are to be completed within 6 weeks prior to registration.
* X-rays and/or scans to determine disease status are to be completed within 6 months prior to registration (or the next business day if falls on a weekend or holiday).

Exclusion Criteria:

* Patients with a prior history of radiation for bladder cancer
* Patients with a prior history of radiation for prostate cancer are eligible for the study
* Greater than or equal to T2N0M0 transitional cell carcinoma of the bladder on current pathology or in the past
* Patients with a prior history of upper tract urothelial carcinoma are eligible for participation in the study as long as there is no evidence of disease for 6 months prior to study enrollment
* Patients with other malignancies are eligible for enrollment in the study but should not be on active treatment for this malignancy within 12 months of study enrollment. Patients with prior history of local treatment for prostate cancer are eligible for participation in the study
* Patients cannot have received Sunitinib or other anti-angiogenic therapy for at least 12 months prior to enrollment in the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BCG and Sunitinib
* Patients with prior systemic infection with BCG are not eligible for the study
* Patients with prior intolerance to BCG may be considered
* Major incisional surgery within 4 weeks of study enrollment
* Bleeding diathesis or unresolved gross hematuria after bladder biopsy
* Known HIV - positive patients may not participate. This is to avoid additional complications that immune suppression and HIV infection may cause due to treatment with BCG, which is a live attenuated bacteria that is known to cause systemic infection in patients who are immunocompromised.
* Patients taking agents that result in immunosuppression are not eligible for the study due to the potential for the increased risk of systemic infection in those patients receiving BCG
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF), cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade 2.
* Patients with history of or who are suspected to have CHF can be included as long as they are asymptomatic and have an ejection fraction that is equal to or above the institutional lower limit of normal by baseline MUGA (obtained within 28 days of registration or the next business day if falls on a weekend or holiday).
* QTc interval > 500 msec on baseline EKG (to be done within 6 weeks prior to registration or the next business day if falls on a weekend or holiday).
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Patient may not have unresolved bacterial infection.
* Patients with hypothyroidism that can not be adequately controlled with medication will be excluded. All patients will be monitored at trial initiation with a TSH.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy.
* All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment.
* Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy.
* The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Weizer, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Mark P. Schoenberg, MD, Baltimore, Maryland
  - Alon Weizer, MD, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Treatment: Intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma.
  Sunitinib: Patients are treated with a 6-week induction course of intravesical bacillus Calmette-Guerin (BCG) followed by a 2 week rest period and 4 week course of oral Sunitinib.
  Patients will receive intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma. Two weeks after completion of BCG, patients will receive Sunitinib (50 mg daily) continuously for 28 days followed by a two week rest period. Patients will be reassessed with transurethral resection and urine cytology. Those with residual/recurrent disease will receive a second course identical to the initial protocol. Those with a complete response following initial or second treatment will be placed on maintenance BCG.
Period: BCG Induction
Arm/Group | Sunitinib Treatment
Started | 43
Completed | 36
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — ineligible | 3
Not completed — noncompliant w. BCG | 1
Not completed — Adverse Event | 1
Period: Beginning Sunitinib Treatment
Arm/Group | Sunitinib Treatment
Started | 36
Completed | 24
Not Completed | 12
Not completed — cystectomy | 5
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Only participants who were able to begin sunitinib treatment were analyzable and therefore are included here.
Arm/Group | Sunitinib Treatment
Number analyzed (Participants) | 36
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [57 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 7
ECOG performance [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living activities of the patient. It goes from 0 to 5, with 0 being no interference with ordinary living and 5 being dead
  Participants
    0 | 33
    1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response at 3 Months
Description: Complete response is defined as no evidence of cancer on bladder biopsy or on a urine test that looks for cancer cells (cytology)
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Treatment
Number analyzed (Participants) | 36
Participants | 26

2. Secondary Outcome: Percentage of Participants Who Experienced a Complete Response at 6 Months, Following Study Regimen.
Description: as for outcome 1
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Treatment
Number analyzed (Participants) | 36
Participants | 27

3. Secondary Outcome: Recurrence-free Survival at 2 Years in Patients With Intact Bladder.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Treatment
Number analyzed (Participants) | 36
percentage of participants | 77 [58 to 88]

4. Secondary Outcome: Number of Participants With Toxicity Related to Treatment With BCG Followed by Sunitinib
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was used to characterize the toxicity: Toxic events are listed by name, body system and grade.
  Note: to fit within character length constraints, "3" below means Grade 3; and S & S means Skin and Subcutaneous system.
Time Frame: 26 months
Population: All participants were followed, by permission, even those who withdrew from full treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Treatment
Number analyzed (Participants) | 36
Participants
  No Toxicity of Grade 3 or higher | 31
  3: Gastrointestinal: febrile diarrhea | 1
  3: Blood and Lymphatic: Thrombocytopenia | 1
  3: S & S: rash on hands, feet | 1
  3: S & S: hand & foot syndrome | 1
  3 S & S: sores on hands & ft; infection: shingles | 1

ADVERSE EVENTS:
Time Frame: 26 months
Groups:
- Sunitinib Treatment: Intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma.
  Sunitinib: Patients are treated with a 6-week induction course of intravesical bacillus Calmette-Guerin (BCG) followed by a 2 week rest period and 4 week course of oral Sunitinib.
  Patients will receive intravesical BCG (81 mg Theracys BCG in 50 ml normal saline) once weekly for 6 weeks within 6 weeks of bladder biopsy confirming high risk non-muscle invasive urothelial carcinoma. Two weeks after completion of BCG, patients will receive Sunitinib (50 mg daily) continuously for 28 days followed by a 2 week rest period. Patients will be reassessed with transurethral resection and urine cytology. Those with residual/recurrent disease will receive a 2nd course identical to the initial protocol. Those with a complete response following initial or second treatment will be placed on maintenance BCG.
Arm/Group | Sunitinib Treatment
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Treatment (N=36)
Rash on Hands/Feet (Skin and subcutaneous tissue disorders) | 1
Hand/Foot Syndrome (Skin and subcutaneous tissue disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
febrile diarrhea (Gastrointestinal disorders) | 1
Sores on Hands/feet (Skin and subcutaneous tissue disorders) | 1
shingles; zoster reactivation (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Treatment (N=36)
Diarrhea (Gastrointestinal disorders) | 12
Hypertension (Vascular disorders) | 16
Thrombocytopenic (Blood and lymphatic system disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 2
Jaundice (Hepatobiliary disorders) | 6
Nausea (Gastrointestinal disorders) | 11
Epislaxis (Respiratory, thoracic and mediastinal disorders) | 2
Lightheadedness (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 21
Edema (General disorders) | 4
Cough (General disorders) | 3
hand and foot pain (General disorders) | 4
Urinary Tract Infection (Infections and infestations) | 6
Sores in mouth (Gastrointestinal disorders) | 9
Gastritis (Gastrointestinal disorders) | 4
Bilirubin increased (Investigations) | 6
Elevated transminases (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Petachiae (Skin and subcutaneous tissue disorders) | 1
Epidymitis (Renal and urinary disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Acid reflux (Gastrointestinal disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Gastrointestinal cramping (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT00794950/Prot_SAP_000.pdf